CLINICAL TRIAL: NCT01686763
Title: Endothelin-1 and Methabolites Concentrations in Mycrodialysis and Cerebrospinal Fluid in Subarachnoid Hemorrhage Patients
Status: Completed | Type: Observational
Sponsor: University of Turin, Italy (Other)
Responsible Party: Principal Investigator, Luciana Mascia, MD, PhD, University of Turin, Italy
Other Study IDs: CEI 1147
Record Dates: First submitted 2012-09-12; First posted 2012-09-18 (Estimated); Last update posted 2013-03-18 (Estimated); Status verified 2009-12

CONDITIONS: Subarachnoid Hemorrhage, Aneurysmal
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- subarachnoid hemorrhage disease: subarachnoid hemorrhage patients

SUMMARY:
Endothelin-1 (ET-1) seems to be involved in the pathogenesis of cerebral vasospasm after subarachnoid hemorrhage. However measurements of cerebrospinal fluid concentrations (CSF) of ET-1 are not sensitive enough to predict the development of vasospasm representing the average value throughout the entire cerebral circulation. Cerebral microdialysis (MD) is a technique able to detect molecule concentrations in a small perivascular area. The investigators performed a prospective observational clinical study to test the hypothesis that MD ET-1 concentrations should be a sensitive predictor for vasospasm.

Patients with subarachnoid hemorrhage at high risk for vasospasm according to Fisher scale admitted to the ICU were consecutively studied. All patients received surgery within 48 hours from the bleeding; MD probe was placed in the area at risk for vasospasm after surgery and samples were hourly collected and analysed to measure lactate, piruvate and glutamate levels; ET-1 levels in CSF and MD fluids were measured from admission until day 7. At admission and after 7 days two angiographies were performed to detect the degree and extent of vasospasm, Transcranial Doppler and neurological evaluation were daily performed. Patients were then classified according to the presence of vasospasm in 3 groups: absence of vasospasm (NV), presence of vasospasm (CV), acute neurological deterioration (AND).

ELIGIBILITY:
Inclusion Criteria:

* diagnosys of subarachnoid hemorrhage
* angiographic proof of aneurysm
* admission within 24 hours from the subarachnoid hemorrhage
* presence of an intraventricular catheter and a microdialysis catheter placed either after admission or at the time of the surgery

Exclusion Criteria:

* moribund
* GCS=3
* denied consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with subarachnoid hemorrhage at high risk for vasospasm according to Fisher scale admitted to the ICU were consecutively studied.
Sampling Method: Non-Probability Sample
Enrollment: 35 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
cerebral vasospasm incidence | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Mascia, MD, PhD, Principal Investigator — University of Turin, Italy